CLINICAL TRIAL: NCT01170130
Title: Efficiency and Safety of Lidocaine Usage for Pupil Dilatation (Mydriasis) During Cataract Surgery
Brief Title: Lidocaine Usage for Pupil Dilatation (Mydriasis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Orna Geyer, professor, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC-09-0017-CTIL
Record Dates: First submitted 2010-07-13; First posted 2010-07-27 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Cataract
Keywords: Cataract; Mydriasis; Lidocaine
MeSH Terms: conditions — Cataract; Mydriasis | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidmyd (Experimental): The same group is used for the first and the second part of the experiment. Initially the patients will be given topical cyclopentolate 1% and Phenylephrine 10% and the pupil diameter will be recorded. In the second part of the experiment lidocaine 1% will be introduced intracamerally and the pupil size will be recorded again. The 2 measurements will be statistically compared/evaluated.
  Interventions: Drug: Lidocaine 1% (sterile)

INTERVENTIONS:
Drug: Lidocaine 1% (sterile) — during the phacoemulsification surgery patients will be given intracamerally lidocaine 1% (0.2 ml) and the pupil size will be recorded after 90 seconds

SUMMARY:
The purpose of this study is to determine if the mydriatic effect of intracameral lidocaine 1% is as effective as topical cyclopentolate 1% and phenylephrine 10% for achieving effective mydriasis during phacoemulsification surgery.

DETAILED DESCRIPTION:
Former studied done on the effect of Intracameral lidocaine 1% compared to topical mydriatic agents for achieving effective mydriasis during phacoemulsification surgery have compared 2 different groups of patients, ie; One group received topical agents and the other received intracameral lidocaine. The resultant pupil size was recorded and evaluated in the 2 groups. Our purpose is to compare the effect of these agents on the same group of people.

Patients recruited will be invited first for evaluation at least 1 week before the surgery. During this evaluation 1 dose (drop) of topical cyclopentolate 1% and Phenylephrine 10% will be instilled to the evaluated eye 3 times at 10 minutes intervals. After 1 hour from the last instillation pupil diameter will be recorded. In the second part of this study during the phacoemulsification surgery patients will be given intracamerally lidocaine 1% (0.2 ml) and the pupil size will be recorded after 90 seconds. the resultant values will be evaluated/compared.

ELIGIBILITY:
Inclusion Criteria:

* cataract
* men and women
* can read and sign informed consent form

Exclusion Criteria:

* sensitivity to Lidocaine
* sensitivity to Ephrine
* any other ocular surgeries
* diseases like Adie's pupil, Horner syndrome

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pupil size after mydriatics | no longer then 1 year
  We would like to evaluate whether Pupil size dilated with Intracameral Lidocaine 1% is as effective dilator compared with Topical Cyclopentolate 1% and Phenylephrine 10%

CONTACTS AND LOCATIONS:
Overall Officials: Orna Geyer, Professor, Principal Investigator — Carmel Medical Center